CLINICAL TRIAL: NCT00749190
Title: A Phase II, Randomized, Parallel Group Safety, Efficacy, and Pharmacokinetics Study of BI 10773 (1 mg, 5 mg, 10 mg, 25 mg, and 50 mg) Administered Orally Once Daily Over 12 Weeks Compared Double Blind to Placebo With an Additional Open-label Sitagliptin Arm in Type 2 Diabetic Patients With Insufficient Glycemic Control Despite Metformin Therapy
Brief Title: BI 10773 add-on to Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1245.10; EudraCT 2008-000641-54
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Sitagliptin Phosphate

INTERVENTIONS:
Drug: BI 10773
Drug: placebo
Drug: sitagliptin

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and pharmacokinetics of five doses of BI 10773 compared to placebo given for 12 weeks as add-on therapy to on going metformin therapy in patients with T2DM with insufficient glycemic control. In addition, there will be an open-label treatment arm with sitagliptin (JanuviaTM) as add-on therapy to metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with a diagnosis of type 2 diabetes mellitus and previously treated with metformin alone or with metformin and one other oral antidiabetic drug
2. Stable metformin therapy of at least 1500 mg/day, or less if that is a maximum tolerated dose.
3. HbA1c at screening 6.5% to 9.0% for patients on metformin and one other antidiabetic drug, and HbA1c >7.0% to 10% for patients on metformin only
4. HbA1c >7.0% to 10.0% at Visit 2 (Start of Run-in)
5. Age >=18 and <80years
6. Body Mass Index (BMI) <=40 kg/m2
7. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

1. Myocardial infarction, stroke or transient ischemic attack (TIA) within 6 months prior to informed consent
2. Impaired hepatic function
3. Renal insufficiency or impaired renal function
4. Diseases of the central nervous system or psychiatric disorders or clinically relevant neurological disorders that may interfere with participation in the trial
5. Chronic or clinically relevant acute infections
6. Current or chronic urogenital tract infection
7. History of clinically relevant allergy/hypersensitivity
8. Treatment with glitazones (e.g., rosiglitazone, pioglitazone), glucagon-like peptide (GLP-1) analogues, or insulin within 3 months prior to informed consent
9. Treatment with anti-obesity drugs within 3 months prior to informed consent
10. Treatment with systemic steroids or change in dosage of thyroid hormones within 6 weeks prior to informed consent
11. Alcohol abuse or drug abuse
12. Treatment with an investigational drug within 2 months prior to informed consent
13. Women of child-bearing potential who are nursing or pregnant, or who are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to periodic pregnancy testing during participation in the trial

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (116):
- United States (19):
  - 1245.10.10026 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1245.10.10001 Boehringer Ingelheim Investigational Site, Mission Viejo, California
  - 1245.10.10011 Boehringer Ingelheim Investigational Site, Pasadena, California
  - 1245.10.10028 Boehringer Ingelheim Investigational Site, Spring Valley, California
  - 1245.10.10027 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 1245.10.10004 Boehringer Ingelheim Investigational Site, Clearwarter, Florida
  - 1245.10.10021 Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - 1245.10.10005 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.10.10019 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1245.10.10024 Boehringer Ingelheim Investigational Site, Saint Cloud, Florida
  - 1245.10.10014 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 1245.10.10016 Boehringer Ingelheim Investigational Site, Staten Island, New York
  - 1245.10.10009 Boehringer Ingelheim Investigational Site, Shelby, North Carolina
  - 1245.10.10006 Boehringer Ingelheim Investigational Site, Wadsworth, Ohio
  - 1245.10.10023 Boehringer Ingelheim Investigational Site, Norristown, Pennsylvania
  - 1245.10.10010 Boehringer Ingelheim Investigational Site, Clemson, South Carolina
  - 1245.10.10015 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.10.10012 Boehringer Ingelheim Investigational Site, Temple, Texas
  - 1245.10.10025 Boehringer Ingelheim Investigational Site, Federal Way, Washington
- Argentina (5):
  - 1245.10.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.10.54004 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.10.54008 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1245.10.54006 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1245.10.54005 Boehringer Ingelheim Investigational Site, Mendoza
- Austria (4):
  - 1245.10.43002 Boehringer Ingelheim Investigational Site, Graz
  - 1245.10.43004 Boehringer Ingelheim Investigational Site, Innsbruck
  - 1245.10.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1245.10.43003 Boehringer Ingelheim Investigational Site, Vienna
- Czechia (4):
  - 1245.10.42003 Boehringer Ingelheim Investigational Site, Brno
  - 1245.10.42005 Boehringer Ingelheim Investigational Site, Brno
  - 1245.10.42001 Boehringer Ingelheim Investigational Site, Břeclav
  - 1245.10.42002 Boehringer Ingelheim Investigational Site, Hodonín
- Estonia (2):
  - 1245.10.37201 Boehringer Ingelheim Investigational Site, Tallinn
  - 1245.10.37202 Boehringer Ingelheim Investigational Site, Tartu
- Finland (4):
  - 1245.10.58006 Boehringer Ingelheim Investigational Site, Kerava
  - 1245.10.58003 Boehringer Ingelheim Investigational Site, Oulu
  - 1245.10.58004 Boehringer Ingelheim Investigational Site, Tampere
  - 1245.10.58001 Boehringer Ingelheim Investigational Site, Turku
- France (28):
  - 1245.10.3302A Boehringer Ingelheim Investigational Site, Bondy
  - 1245.10.3302B Boehringer Ingelheim Investigational Site, Bondy
  - 1245.10.3310A Boehringer Ingelheim Investigational Site, Caen
  - 1245.10.3310B Boehringer Ingelheim Investigational Site, Caen
  - 1245.10.3310C Boehringer Ingelheim Investigational Site, Caen
  - 1245.10.3301A Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - 1245.10.3301B Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - 1245.10.3303A Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.10.3303B Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.10.3303C Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.10.3303D Boehringer Ingelheim Investigational Site, La Rochelle
  - 1245.10.3308A Boehringer Ingelheim Investigational Site, Le Grau-du-Roi
  - 1245.10.3308B Boehringer Ingelheim Investigational Site, Le Grau-du-Roi
  - 1245.10.3309A Boehringer Ingelheim Investigational Site, Nanterre
  - 1245.10.3306A Boehringer Ingelheim Investigational Site, Narbonne
  - 1245.10.3306B Boehringer Ingelheim Investigational Site, Narbonne
  - 1245.10.3307A Boehringer Ingelheim Investigational Site, Quimper
  - 1245.10.3304A Boehringer Ingelheim Investigational Site, Reims
  - 1245.10.3304B Boehringer Ingelheim Investigational Site, Reims
  - 1245.10.3304C Boehringer Ingelheim Investigational Site, Reims
  - 1245.10.3311A Boehringer Ingelheim Investigational Site, Saint-Mandé
  - 1245.10.3311B Boehringer Ingelheim Investigational Site, Saint-Mandé
  - 1245.10.3311C Boehringer Ingelheim Investigational Site, Saint-Mandé
  - 1245.10.3311D Boehringer Ingelheim Investigational Site, Saint-Mandé
  - 1245.10.3305A Boehringer Ingelheim Investigational Site, Valenciennes
  - 1245.10.3305B Boehringer Ingelheim Investigational Site, Valenciennes
  - 1245.10.3305C Boehringer Ingelheim Investigational Site, Valenciennes
  - 1245.10.3305D Boehringer Ingelheim Investigational Site, Valenciennes
- Germany (4):
  - 1245.10.49001 Boehringer Ingelheim Investigational Site, Erlangen
  - 1245.10.49003 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1245.10.49002 Boehringer Ingelheim Investigational Site, Hamburg
  - 1245.10.49004 Boehringer Ingelheim Investigational Site, Rehlingen-Siersburg
- Hungary (5):
  - 1245.10.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.10.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.10.36004 Boehringer Ingelheim Investigational Site, Budapest
  - 1245.10.36005 Boehringer Ingelheim Investigational Site, Győr
  - 1245.10.36002 Boehringer Ingelheim Investigational Site, Szombathely
- Latvia (7):
  - 1245.10.37101 Boehringer Ingelheim Investigational Site, Daugavpils
  - 1245.10.37105 Boehringer Ingelheim Investigational Site, Kuldīga
  - 1245.10.37106 Boehringer Ingelheim Investigational Site, Ogre
  - 1245.10.37103 Boehringer Ingelheim Investigational Site, Riga
  - 1245.10.37107 Boehringer Ingelheim Investigational Site, Riga
  - 1245.10.37102 Boehringer Ingelheim Investigational Site, Talsi
  - 1245.10.37104 Boehringer Ingelheim Investigational Site, Valmiera
- Norway (4):
  - 1245.10.47004 Boehringer Ingelheim Investigational Site, Ålesund
  - 1245.10.47003 Boehringer Ingelheim Investigational Site, Hamar
  - 1245.10.47005 Boehringer Ingelheim Investigational Site, Oslo
  - 1245.10.47001 Boehringer Ingelheim Investigational Site, Stavanger
- Romania (7):
  - 1245.10.40001 Boehringer Ingelheim Investigational Site, Alba Iulia
  - 1245.10.40005 Boehringer Ingelheim Investigational Site, Baia Mare Maramures
  - 1245.10.40003 Boehringer Ingelheim Investigational Site, Brasov
  - 1245.10.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1245.10.40007 Boehringer Ingelheim Investigational Site, Bucharest
  - 1245.10.40004 Boehringer Ingelheim Investigational Site, Galati
  - 1245.10.40006 Boehringer Ingelheim Investigational Site, Satu Mare
- Russia (7):
  - 1245.10.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.10.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.10.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.10.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.10.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.10.70006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.10.70007 Boehringer Ingelheim Investigational Site, Saratov
- Slovakia (4):
  - 1245.10.62003 Boehringer Ingelheim Investigational Site, Bratislava
  - 1245.10.62001 Boehringer Ingelheim Investigational Site, Nitra
  - 1245.10.62002 Boehringer Ingelheim Investigational Site, Nitra
  - 1245.10.62004 Boehringer Ingelheim Investigational Site, Prešov
- Spain (7):
  - 1245.10.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1245.10.34001 Boehringer Ingelheim Investigational Site, Girona
  - 1245.10.34010 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1245.10.34004 Boehringer Ingelheim Investigational Site, Málaga
  - 1245.10.34005 Boehringer Ingelheim Investigational Site, Palma (Mallorca)
  - 1245.10.34006 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1245.10.34008 Boehringer Ingelheim Investigational Site, Santander
- Ukraine (5):
  - 1245.10.38002 Boehringer Ingelheim Investigational Site, Dnipro
  - 1245.10.38004 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.10.38005 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.10.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.10.38001 Boehringer Ingelheim Investigational Site, Vinnitsa

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Riggs MM, Staab A, Seman L, MacGregor TR, Bergsma TT, Gastonguay MR, Macha S. Population pharmacokinetics of empagliflozin, a sodium glucose cotransporter 2 inhibitor, in patients with type 2 diabetes. J Clin Pharmacol. 2013 Oct;53(10):1028-38. doi: 10.1002/jcph.147. Epub 2013 Aug 13. PMID 23940010

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients receive Placebo in tablets matching the Empagliflozin tablets in appearance once daily.
- Empagliflozin 1 mg: Patients receive 1 mg Empagliflozin in tablets once daily.
- Empagliflozin 5 mg: Patients receive 5 mg Empagliflozin in tablets once daily.
- Empagliflozin 10 mg: Patients receive 10 mg Empagliflozin in tablets once daily.
- Empagliflozin 25 mg: Patients receive 25 mg Empagliflozin in tablets once daily.
- Empagliflozin 50 mg: Patients receive 50 mg Empagliflozin in tablets once daily.
- Sitagliptin OL: Patients receive 100 mg Sitagliptin (open-label) in tablets once daily.
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Started | 71 | 71 | 71 | 71 | 70 | 70 | 71
Completed | 66 | 66 | 70 | 66 | 70 | 65 | 70
Not Completed | 5 | 5 | 1 | 5 | 0 | 5 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 4 | 0 | 3 | 0
Not completed — Lack of Efficacy | 3 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Other reason not defined above | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) consisting of all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Empa 1 mg: Patients receive 1 mg Empagliflozin in tablets once daily.
- Empa 5 mg: Patients receive 5 mg Empagliflozin in tablets once daily.
- Empa 10 mg: Patients receive 10 mg Empagliflozin in tablets once daily.
- Empa 25 mg: Patients receive 25 mg Empagliflozin in tablets once daily.
- Empa 50 mg: Patients receive 50 mg Empagliflozin in tablets once daily.
- Sitag: Patients receive 100 mg Sitagliptin (open-label) in tablets once daily.
- Total: Total of all reporting groups
Arm/Group | Placebo | Empa 1 mg | Empa 5 mg | Empa 10 mg | Empa 25 mg | Empa 50 mg | Sitag | Total
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 70 | 70 | 71 | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.5) | 57.4 (8.8) | 59.7 (7.3) | 59.0 (9.0) | 58.7 (8.1) | 55.9 (9.4) | 57.6 (10.1) | 58.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 30 | 42 | 38 | 33 | 31 | 33 | 245
  Male | 33 | 41 | 29 | 33 | 37 | 39 | 38 | 250

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c After 12 Weeks of Treatment
Description: Change from baseline in HbA1c after 12 weeks of treatment.
  In the measured values adjusted means are displayed. For means for the placebo and empagliflozin arms are from the model excluding the sitagliptin open label (OL) arm. The mean for the sitagliptin OL arm is from the model with just this treatment group and the placebo group.
Time Frame: Baseline and 12 weeks
Population: Full analysis set (FAS) consisting of all randomized patients who were treated with at least one dose of study drug and has a baseline measurement of the primary endpoint. The imputation method used was a modified last observation carried forward (LOCF) approach which used linear interpolation, LOCF and worst observation carried forward (WOCF).
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 70 | 70 | 71
percentage of HbA1c | 0.15 (0.08) | -0.09 (0.08) | -0.23 (0.08) | -0.56 (0.08) | -0.55 (0.08) | -0.49 (0.08) | -0.45 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 1 mg; Test type: Superiority or Other; p = 0.0226, ANCOVA — P-values are regarded as descriptive, adjustment for multiple testing was not necessary; Based on ANCOVA with terms for treatment, number of previously used anti-diabetic medications, country and baseline; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.44 to -0.03], Standard Error of Mean 0.10 — Difference calculated as empagliflozin 1 mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 5 mg; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-values are regarded as descriptive, adjustment for multiple testing was not necessary; Based on ANCOVA with terms for treatment, number of previously used anti-diabetic medications, country and baseline; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.59 to -0.18], Standard Error of Mean 0.10 — Difference calculated as empagliflozin 5 mg minus placebo
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values are regarded as descriptive, adjustment for multiple testing was not necessary; Based on ANCOVA with terms for treatment, number of previously used anti-diabetic medications, country and baseline; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-0.91 to -0.51], Standard Error of Mean 0.10 — Difference calculated as empagliflozin 10 mg minus placebo
Statistical Analysis 4: Comparison: Placebo vs Empagliflozin 25 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values are regarded as descriptive, adjustment for multiple testing was not necessary; Based on ANCOVA with terms for treatment, number of previously used anti-diabetic medications, country and baseline; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-0.91 to -0.50], Standard Error of Mean 0.10 — Difference calculated as empagliflozin 25 mg minus placebo
Statistical Analysis 5: Comparison: Placebo vs Empagliflozin 50 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values are regarded as descriptive, adjustment for multiple testing was not necessary; Based on ANCOVA with terms for treatment, number of previously used anti-diabetic medications, country and baseline; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-0.84 to -0.43], Standard Error of Mean 0.10 — Difference calculated as empagliflozin 50 mg minus placebo

2. Secondary Outcome: Change of FPG From Baseline After 12 Weeks of Treatment
Description: Change of Fasting Plasma Glucose (FPG) from baseline after 12 weeks of treatment. Results presented stem from a repeated measures analysis.
  In the measured values adjusted means are displayed. For means for the placebo and empagliflozin arms are from the model excluding the sitagliptin open label (OL) arm. The mean for the sitagliptin OL arm is from the model with just this treatment group and the placebo group.
Time Frame: Baseline and 12 weeks
Population: FAS using modified LOCF imputation method
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 69 | 68 | 70 | 68 | 69 | 69 | 69
mg/dL | 4.75 (3.48) | -1.70 (3.49) | -15.84 (3.45) | -22.14 (3.49) | -26.83 (3.47) | -27.91 (3.47) | -12.92 (4.73)

3. Secondary Outcome: Change of HbA1c From Baseline Over Time
Description: Change of HbA1c from baseline over time. Results presented stem from a repeated measures analysis.
Time Frame: Baseline and weeks 4, 8 and 12
Population: FAS. Imputation method used was the classical LOCF (CLOCF) approach which uses always the last available value.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 70 | 70 | 71
percentage of HbA1c
  Week 4 | 0.02 (0.06) | -0.12 (0.06) | -0.16 (0.06) | -0.32 (0.06) | -0.31 (0.06) | -0.36 (0.06) | -0.26 (0.06)
  Week 8 | 0.05 (0.07) | -0.14 (0.07) | -0.30 (0.07) | -0.57 (0.07) | -0.52 (0.07) | -0.53 (0.07) | -0.40 (0.07)
  Week 12 | 0.12 (0.08) | -0.08 (0.08) | -0.27 (0.08) | -0.57 (0.08) | -0.59 (0.08) | -0.50 (0.08) | -0.45 (0.08)

4. Secondary Outcome: Proportion of Patients Who Achieve an HbA1c ≤7.0% After 12 Weeks of Treatment
Description: Results for HbA1c categories at week 12 (Proportion of patients with HbA1c less than equal to 7%) based on logistic regression
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 70 | 70 | 71
percentage of participants | 15.5 | 23.9 | 21.1 | 38.0 | 37.1 | 35.7 | 33.8

5. Secondary Outcome: Proportion of Patients Who Achieve an HbA1c Lowering of at Least 0.5% After 12 Weeks of Treatment
Description: Results for HbA1c categories at week 12 (Proportion of patients with HbA1c lowered at least 0.5%) based on logistic regression
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 70 | 70 | 71
percentage of participants | 21.1 | 31.0 | 40.8 | 60.6 | 60.0 | 48.6 | 53.5

6. Secondary Outcome: Change From Baseline to Week 12 in Fasting Plasma Insulin (FPI)
Description: Results for change of FPI from baseline at week 12 based on ANCOVA
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Mean (Standard Error); unit: mU/L
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 63 | 59 | 60 | 59 | 57 | 61 | 59
mU/L | 0.43 (0.57) | 0.09 (0.59) | -0.84 (0.58) | -1.77 (0.58) | -0.11 (0.59) | -1.52 (0.57) | 1.84 (0.58)

7. Secondary Outcome: Change in Homeostasis Model Assessment Index for Insulin Resistance (HOMA-IR)
Description: HOMA-IR (to assess insulin resistance) is defined as (FPI x FPG)/22.5. Results based on ANCOVA.
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Mean (Standard Error); unit: mU/L x mmol/L
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 62 | 58 | 59 | 59 | 57 | 59 | 59
mU/L x mmol/L | 0.23 (0.26) | -0.11 (0.27) | -0.60 (0.26) | -1.04 (0.26) | -0.52 (0.27) | -1.10 (0.27) | 0.48 (0.26)

8. Secondary Outcome: Change in Homeostasis Model Assessment Index for Beta Cell Function (HOMA-%B)
Description: HOMA-%B (to assess insulin beta cell function) is defined as (20 x FPI)/(FPG-3.5), FPG in mg/dl. Results are based on ANCOVA.
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Mean (Standard Error); unit: mU / mmol
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 62 | 58 | 58 | 59 | 57 | 59 | 59
mU / mmol | 0.30 (2.70) | 0.08 (2.77) | 0.36 (2.76) | 1.55 (2.72) | 6.68 (2.78) | 4.01 (2.76) | 12.38 (2.75)

9. Secondary Outcome: Change of Body Weight After 12 Weeks of Treatment
Description: Results for change of body weight after 12 weeks of treatment based on ANCOVA.
Time Frame: Baseline and 12 weeks
Population: FAS (CLOCF)
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Number analyzed (Participants) | 71 | 71 | 71 | 71 | 70 | 70 | 71
kg | -1.16 (0.31) | -1.55 (0.31) | -2.28 (0.31) | -2.74 (0.31) | -2.56 (0.31) | -2.85 (0.32) | -0.84 (0.31)

10. Secondary Outcome: Trough Concentrations of Empagliflozin in Plasma
Description: (Pre-dose) trough concentrations of Empagliflozin in plasma, within 30 minutes of dosing.
Time Frame: Days 28, 56 and 84
Population: All patients who received at least one dose of Empagliflozin and have some Pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg
Number analyzed (Participants) | 58 | 65 | 64 | 61 | 63
nmol/L
  Day 28 (N=58, 65, 62, 58, 63) | 3.19 (88.8) | 13.1 (79.4) | 27.3 (127) | 92.5 (111) | 119 (78.7)
  Day 56 (N=56, 64, 64, 61, 61) | 2.93 (69.6) | 11.5 (63.2) | 23.0 (93.8) | 75.4 (140) | 119 (85.5)
  Day 84 (N=53, 61, 59, 57, 57) | 2.87 (80.1) | 11.2 (69.6) | 23.4 (85.1) | 71.0 (111) | 112 (79.6)

ADVERSE EVENTS:
Time Frame: From first dose of study medication until 7 days following the last intake of study medication, up to 100 days
Arm/Group | Placebo | Empagliflozin 1 mg | Empagliflozin 5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Empagliflozin 50 mg | Sitagliptin OL
Serious Adverse Events (participants affected / at risk) | 2/71 | 0/71 | 3/71 | 1/71 | 2/70 | 3/70 | 0/71
Other Adverse Events (participants affected / at risk) | 4/71 | 2/71 | 2/71 | 7/71 | 4/70 | 3/70 | 4/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Empagliflozin 1 mg (N=71) | Empagliflozin 5 mg (N=71) | Empagliflozin 10 mg (N=71) | Empagliflozin 25 mg (N=70) | Empagliflozin 50 mg (N=70) | Sitagliptin OL (N=71)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Empagliflozin 1 mg (N=71) | Empagliflozin 5 mg (N=71) | Empagliflozin 10 mg (N=71) | Empagliflozin 25 mg (N=70) | Empagliflozin 50 mg (N=70) | Sitagliptin OL (N=71)
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 3 | 4 | 1 | 2
Hypertension (Vascular disorders) | 2 | 0 | 1 | 4 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.